CLINICAL TRIAL: NCT06393205
Title: Efficacy of Naso-Esophageal Tube Feeding in Patients With High Cervical Spinal Cord Injury: A Randomized Controlled Study
Brief Title: Efficacy of Naso-Esophageal Tube Feeding in Patients With High Cervical Spinal Cord Injury.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Bi shidao
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injury Cervical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Naso-Esophageal Tube Feeding group (Experimental): The patients will be given Naso-Esophageal Tube Feeding and routine treatment, for 15 days.
  Interventions: Device: Naso-Esophageal Tube Feeding; Behavioral: Routine treatment
- The Nasogastric Tube Feeding group (Active Comparator): The patients will be given Nasogastric Tube Feeding and routine treatment, for 15 days.
  Interventions: Device: Nasogastric Tube Feeding; Behavioral: Routine treatment

INTERVENTIONS:
Device: Naso-Esophageal Tube Feeding — During nasogastric tube feeding, a thin, flexible tube is carefully inserted through one nostril and passed down the throat into the stomach. Once in place, liquid nutrition, medication, or fluids can be administered through the tube, providing essential nutrients and hydration directly to the patient's digestive system. Nasogastric tube feeding may be used temporarily to support patients during acute illness or surgery, or it may be a long-term solution for individuals with chronic conditions that affect their ability to eat normally.
  Arms: the Naso-Esophageal Tube Feeding group
Device: Nasogastric Tube Feeding — The control group was given enteral nutritional support with Nasogastric Tube Feeding according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the patient cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements. The feeding content was formulated by the nutritionists based on the patients condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups. For patients with limited tube feeding compliance, we made appropriate adjustments to ensure that they were not at risk of severe malnutrition as much as possible.
  Arms: The Nasogastric Tube Feeding group
Behavioral: Routine treatment — Including： Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.

SUMMARY:
The goal of this clinical trial is to compare the differences in Pneumonia situation and nutritional status between Patients With High Cervical Spinal Cord Injury using Naso-Esophageal Tube Feeding and Nasogastric Tube. Patients will be randomly divided into an observation group and a control group, all receiving routine rehabilitation treatment. On this basis, the observation group will use Naso-Esophageal Tube Feeding for enteral nutrition support, while the control group will use Nasogastric Tube. Researchers will compare changes in Pneumonia situation and nutritional status of two groups of patients before and after the study to see if Naso-Esophageal Tube Feeding can improve the Pneumonia situation and nutritional status between Patients With High Cervical Spinal Cord Injury

DETAILED DESCRIPTION:
Naso-esophageal tube feeding is a medical procedure utilized to provide nutrition directly into the esophagus via a tube inserted through the nose. This method is employed when individuals cannot consume food orally due to various medical conditions, such as dysphagia (difficulty swallowing), neurological disorders, or conditions affecting the upper gastrointestinal tract.

The goal of this clinical trial is to compare the differences in Pneumonia situation and nutritional status between Patients With High Cervical Spinal Cord Injury using Naso-Esophageal Tube Feeding and Nasogastric Tube. Patients will be randomly divided into an observation group and a control group, all receiving routine rehabilitation treatment. On this basis, the observation group will use Naso-Esophageal Tube Feeding for enteral nutrition support, while the control group will use Nasogastric Tube. Researchers will compare changes in Pneumonia situation and nutritional status of two groups of patients before and after the study to see if Naso-Esophageal Tube Feeding can improve the Pneumonia situation and nutritional status between Patients With High Cervical Spinal Cord Injury

ELIGIBILITY:
Inclusion Criteria:

* High Cervical Spinal Cord Injury.
* any degree of dysphagia at admission;
* steady vital signs, without severe cognitive impairment or sensory aphasia, able to cooperate with the assessment.

Exclusion Criteria:

* damaged mucosa or incomplete structure in nasopharynx;
* unfeasible to the support of parenteral nutrition;
* simultaneously suffering from liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Nutritional status-total protein | Day 1 and day 15
  The relevant indicators include total protein (TP, g/L) from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.
Nutritional status-hemoglobin | Day 1 and day 15
  The relevant indicators include hemoglobin (Hb, g/L)from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.
Nutritional status-albumin | Day 1 and day 15
  The relevant indicators include albumin (ALB, g/L)from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.
Nutritional status-prealbumin | Day 1 and day 15
  The relevant indicators include prealbumin (PA, mg/L) from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.

SECONDARY OUTCOMES:
Body weight | Day 1 and day 15
  Body weight measurement of the infants was conducted by the same nurse according to the relevant standards.
Swallowing Quality of Life questionnaire | Day 1 and day 15
  Swallowing Quality of Life questionnaire was used to evaluate the quality of life, which consists of 44 items and divided into 11 main domains, including: overall satisfaction, understanding, diet, hydration, communication, respiratory issues, postoperative recovery, social impact, mental health, saliva control, and appearance. The maximum rough score was 220 points, which was converted into a standard percentage system in our study. As the scores increased, the quality of life was better.
Dysphagia Handicap Index | Day 1 and day 15
  Dysphagia Handicap Index is a self-reported questionnaire used to assess the impact of dysphagia on an individual's quality of life. It typically consists of multiple questions related to the physical, functional, and emotional aspects of swallowing difficulties. The total score range varies between 0 and 100. A higher score indicates a greater perceived impact of dysphagia on the individual's quality of life.
Pneumonia | Day 1 and day 15
  The occurrence of pneumonia in patients was assessed before and after treatment. Specifically, first of all, the symptom assessment and physical examination were conducted to all patients, during which, the doctor would inquire symptoms related to pneumonia, such as cough, sputum production, difficulty breathing, chest pain, etc. and observe the patient's respiratory condition, including respiratory rate, breath sounds, and any abnormal signs in the chest.